CLINICAL TRIAL: NCT06027372
Title: Differences in Heart Rate Variability and Nocturnal Blood Oxygen Saturation of Patients With Idiopathic Pulmonary Fibrosis Between at Baseline and During Acute Exacerbation
Brief Title: Heart Rate Variability and Nocturnal Blood Oxygen Saturation in Patients With Idiopathic Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-04-016BC
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPF patients with acute exacerbation during test period: IPF patients completing pulmonary function, overnight SpO2 monitor and "LARGAN" ECG Holter reqire hospitalization during test period.
  Interventions: Device: "LARGAN" ECG Holter
- IPF patients without acute exacerbation during test period: IPF patients completing pulmonary function, overnight SpO2 monitor and "LARGAN" ECG Holter remain stable during test period.
  Interventions: Device: "LARGAN" ECG Holter

INTERVENTIONS:
Device: "LARGAN" ECG Holter — wear "LARGAN" ECG Holter during sleep once after completion of pulmonary function test

SUMMARY:
The goal of this observational study is to compare the overnight heart rate variability (HRV) and nocturnal oxygen saturation (SpO2) in patients with idiopathic pulmonary fibrosis (IPF). The main questions it aims to answer are: (1). if there are correlations between pulmonary function test and HRV and overnight SpO2; (2). if HRV and SpO2 can predict the occurrence of acute exacerbation in patients with IPF. Participants will be asked to examine pulmonary function test (including lung volumes and six-minute walk test) and wear pulse oxygenation recorder and "LARGAN" ECG Holter" ("LARGAN HEALTH TECHNOLOGY" Sleep Apnea And Sleep Quality Examination System) during sleep.

ELIGIBILITY:
Inclusion Criteria:

* individuals meet the diagnosis of idiopathic pulmonary fibrosis
* individuals agree to participate this study and sign the informed consent
* individuals have cognitive and behavioral abilities

Exclusion Criteria:

* age less than 50 years old
* individuals refuse to participate this study and sign the informed consent
* individuals of unclear consciousness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals meet the diagnosis of idiopathic pulmonary fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-08-27 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The correlations between measures of pulmonary function test and heart rate variability | 1 day test duration

CONTACTS AND LOCATIONS:
Overall Officials: Diahn-Warng Perng, PhD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
under reasonable request